CLINICAL TRIAL: NCT01621594
Title: Prospective Evaluation of New Techniques in Radiation Reduction for Cardiovascular Computed Tomographic Angiography
Brief Title: Evaluating New Radiation Techniques for Cardiovascular Imaging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 120141; 12-H-0141
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2025-12-12

CONDITIONS: Coronary Disease
Keywords: computer tomography; Cardiac; Radiation Reduction; Iterative Reconstruction
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Subjects with Clinical indication for a coronary CT angiography exam
  Interventions: Device: Cannon Aquilion ONE CT system

INTERVENTIONS:
Device: Cannon Aquilion ONE CT system — To test the diagnostic accuracy of low-radiation dose CT coronary angiography for detecting significant coronary artery stenosis and to determine the prognostic value of low-radiation dose CT coronary angiography for discriminating patient risk of death or major adverse cardiac events.

SUMMARY:
Title: Evaluating New Radiation Techniques for Cardiovascular Imaging

Background:

Cardiac CT angiography is associated with radiation exposure. Different methods of creating CT pictures have been developed to reduce the radiation dose to the subject. The purpose of this research study is to learn whether these low dose research imagings are accurate or predict subject outcomes.

Cardiac CT is also used for diagnostic imaging of coronary artery disease and identification of abnormal cardiac structures. An additional purpose of this study is to monitor the progression of cardiac disease.

Cardiac imaging software and AI are constantly evolving and requires validation for accuracy. Using existing scan data, updated image software reconstruction can be applied and compared to previous existing standard of care images.

Objectives:

- To study new ways of taking pictures of the heart or blood vessels using computed tomography.

Eligibility:

- Adults at least 18 years of age who will be having imaging studies to help detect heart or blood vessel problems.

Design:

* Participants will be screened with a physical exam and medical history. Blood samples will be taken to check kidney function.
* Participants will have a CT scan of the heart and blood vessels. A contrast agent may be used to improve the quality of the images. The scanning session may last up to 2 hours.
* Timing of and the need for follow up contact will depend on results from the initial scan and may be repeated to assess for late events. Telephone, office contact, or other follow-up of subjects may be done after CCTA to evaluate if the subject had subsequent cardiovascular testing. Further follow up will be based on reported test results.

DETAILED DESCRIPTION:
Cardiac CT angiography is associated with radiation exposure. Different methods of creating CT pictures have been developed to reduce the radiation dose to the subject. The purpose of this research study is to learn whether these low dose research imagings are accurate or predict subject outcomes.

Cardiac CT is also used for diagnostic imaging of coronary artery disease and identification of abnormal cardiac structures. An additional purpose of this study is to monitor the progression of cardiac disease.

Cardiac imaging software and Artificial Intelligence (AI) are constantly evolving and requires validation for accuracy. Using existing scan data, updated image software reconstruction can be applied and compared to previous existing standard of care images.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Clinical indication for a coronary CT angiography exam
  2. Age equal to or greater than 18 years
  3. Able to understand and willing to sign the Informed Consent Form
  4. Able and willing to provide follow-up information

EXCLUSION CRITERIA:

1. Pregnancy
2. If receiving intravenous contrast, severe renal excretory dysfunction, estimated glomerular filtration rate < 30 mL/min/1.73m2 body surface area according to the Modification of Diet in Renal Disease criteria or as reported by the clinical lab. Glomerular filtration rate will be estimated using the 2021 CK-EPI equation that eliminate the use of race coefficient as reported in CRIS.

Screen Failures: Subjects who are screen failures can be re-enrolled once they meet eligibility criteria. Rescreened participants will be assigned the same participant number as for the initial screening.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2012-06-21 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Compare time-to-first cardiovascular events (death, revascularization more than 90 days after CTA, hospitalization, non-fatal myocardial infarction, stroke) in subjects with >=50% coronary stenosis vs. <50% stenosis. | ongoing
  The purpose of this research study is to learn whether these new imaging methods are accurate or predict subject outcomes.

SECONDARY OUTCOMES:
Compare and/or validate radiation saving techniques such as iterative reconstruction or artificial intelligence based methods against standard imaging techniques for calcium scoring. | ongoing
  The purpose of this research study is to learn whether these new imaging methods are accurate or predict subject outcomes.
Evaluate natural history of coronary plaques in subjects with serial imaging if requested by ordering physician, or in subjects with >50% stenosis or high risk plaques on medical therapy. | ongoing
  The purpose of this research study is to learn whether these new imaging methods are accurate or predict subject outcomes.
Estimate diagnostic accuracy of cardiovascular evaluations using current CT technology vs. invasive angiography reports/images and vs. stress perfusion MRI reports/images. | ongoing
  The purpose of this research study is to learn whether these new imaging methods are accurate or predict subject outcomes.
Evaluate image quality from new CT technology. | ongoing
  The purpose of this research study is to learn whether these new imaging methods are accurate or predict subject outcomes.
Survival analysis of subjects identified by CT with significant coronary artery disease (=50% stenosis) vs. subjects without significant coronary artery disease (<50% stenosis). | ongoing
  The purpose of this research study is to learn whether these new imaging methods are accurate or predict subject outcomes.
Estimate radiation dose from clinically performed cardiovascular CT at the NIH compared to outside clinically indicated CTs. | ongoing
  The purpose of this research study is to learn whether these new imaging methods are accurate or predict subject outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Y Chen, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sorokin AV, Hong CG, Aponte AM, Florida EM, Tang J, Patel N, Baranova IN, Li H, Parel PM, Chen V, Wilson SR, Ongstad EL, Collen A, Playford MP, Eggerman TL, Chen MY, Kotani K, Bocharov AV, Remaley AT. Association of oxidized ApoB and oxidized ApoA-I with high-risk coronary plaque features in cardiovascular disease. JCI Insight. 2023 Oct 23;8(20):e172893. doi: 10.1172/jci.insight.172893. PMID 37698922
- [Derived] Sato M, Neufeld EB, Playford MP, Lei Y, Sorokin AV, Aponte AM, Freeman LA, Gordon SM, Dey AK, Jeiran K, Hamasaki M, Sampson ML, Shamburek RD, Tang J, Chen MY, Kotani K, Anderson JL, Dullaart RP, Mehta NN, Tietge UJ, Remaley AT. Cell-free, high-density lipoprotein-specific phospholipid efflux assay predicts incident cardiovascular disease. J Clin Invest. 2023 Sep 15;133(18):e165370. doi: 10.1172/JCI165370. PMID 37471145
- [Derived] Sorokin AV, Patel N, Abdelrahman KM, Ling C, Reimund M, Graziano G, Sampson M, Playford MP, Dey AK, Reddy A, Teague HL, Stagliano M, Amar M, Chen MY, Mehta NN, Remaley AT. Complex association of apolipoprotein E-containing HDL with coronary artery disease burden in cardiovascular disease. JCI Insight. 2022 May 23;7(10):e159577. doi: 10.1172/jci.insight.159577. PMID 35389891
- [Derived] Choi AD, Leifer ES, Yu J, Shanbhag SM, Bronson K, Arai AE, Chen MY. Prospective evaluation of the influence of iterative reconstruction on the reproducibility of coronary calcium quantification in reduced radiation dose 320 detector row CT. J Cardiovasc Comput Tomogr. 2016 Sep-Oct;10(5):359-63. doi: 10.1016/j.jcct.2016.07.016. Epub 2016 Jul 27. PMID 27591767
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2012-H-0141.html